CLINICAL TRIAL: NCT03758937
Title: Comparison of Volume Controlled Ventilation and Pressure Controlled Ventilation in Terms of Respiratory Mechanics in Laparoscopic Bariatric Surgery
Brief Title: Comparison of Volume Controlled Ventilation and Pressure Controlled Ventilation in Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AntalyaTRH31
Record Dates: First submitted 2018-11-27; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Bariatric Surgery
Keywords: bariatric surgery; volume-controlled ventilation; pressure-controlled ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- volume-controlled ventilation group (Active Comparator): During the operation, necessary interventions were made by following the algorithm. Hemodynamic and mechanical ventilation parameters of patients were recorded 5 minutes after induction, 30 minutes after pneumoperitoneum and at the end of surgery and were performed arterial blood gas analysis.
  Interventions: Procedure: volume-controlled ventilation
- pressure-controlled ventilation group (Active Comparator): During the operation, necessary interventions were made by following the algorithm. Hemodynamic and mechanical ventilation parameters of patients were recorded 5 minutes after induction, 30 minutes after pneumoperitoneum and at the end of surgery and were performed arterial blood gas analysis.
  Interventions: Procedure: pressure-controlled ventilation

INTERVENTIONS:
Procedure: volume-controlled ventilation
  Arms: volume-controlled ventilation group
Procedure: pressure-controlled ventilation
  Arms: pressure-controlled ventilation group

SUMMARY:
The purpose of this study is to compare volume controlled-ventilation (VCV) and pressure-controlled ventilation (PCV) in terms of pulmonary gas exchange, respiratory mechanics and arterial blood gas values in patients undergoing laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
Today, morbid obesity has become a global problem. It is not clear which mechanical ventilation mode will be used in bariatric surgery, which is one of the treatment options of these patients. VCV is the most commonly used mode to ventilate anesthetized patients. However, especially in obese patients, high airway pressures and hypoxia may occur due to increased intrapulmonary shunts. Therefore, we aimed to investigate the potential of PCV strategy to improve pulmonary gas exchange, respiratory mechanics and arterial blood gas values according to VCV in patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above,
* ASA II patients
* BMI > 40 kg / m2
* No serious comorbidity.

Exclusion Criteria:

* Unstable patients during the operation
* The requirement for mechanical ventilation in the postoperative period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Partial oxygen pressure | 5 minutes after induction
  Assessed 5 minutes after induction by using arterial blood gas analysis.
Partial oxygen pressure | 30 minutes after pneumoperitoneum
  Assessed 30 minutes after pneumoperitoneum by using arterial blood gas
Partial oxygen pressure | through surgery completion, an average of 90 minutes
  Assessed through surgery completion, an average of 90 minutes by using arterial blood gas

SECONDARY OUTCOMES:
Partial carbon dioxide pressure | 5 minutes after induction, 30 minutes after pneumoperitoneum, through surgery completion, an average of 90 minutes
  Assessed 5 minutes after induction, 30 minutes after pneumoperitoneum and through surgery completion, an average of 90 minutes by using arterial blood gas analysis.
Partial carbon dioxide pressure - end-tidal carbon dioxide pressure | 5 minutes after induction, 30 minutes after pneumoperitoneum, through surgery completion, an average of 90 minutes
  Assessed 5 minutes after induction, 30 minutes after pneumoperitoneum and through surgery completion, an average of 90 minutes by using arterial blood gas analysis and end-tidal monitor.
Peak airway pressure | 5 minutes after induction, 30 minutes after pneumoperitoneum, through surgery completion, an average of 90 minutes
  Assessed 5 minutes after induction, 30 minutes after pneumoperitoneum and through surgery completion, an average of 90 minutes by using the patient monitor.
Dynamic compliance | 5 minutes after induction, 30 minutes after pneumoperitoneum, through surgery completion, an average of 90 minutes
  Assessed 5 minutes after induction, 30 minutes after pneumoperitoneum and through surgery completion, an average of 90 minutes by using formula (Tidal volume/peak airway pressure - Positive end-expiratory pressure)
Inspired oxygen pressure / Fractional oxygen ratio | 5 minutes after induction, 30 minutes after pneumoperitoneum, through surgery completion, an average of 90 minutes
  Assessed 5 minutes after induction, 30 minutes after pneumoperitoneum and through surgery completion, an average of 90 minutes
Alveolar-arterial oxygen gradient pressure | 5 minutes after induction, 30 minutes after pneumoperitoneum, through surgery completion, an average of 90 minutes
  Assessed 5 minutes after induction, 30 minutes after pneumoperitoneum and through surgery completion, an average of 90 minutes by using formula (D(A-a) O2).

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Ozyurt, MD, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Traning and Research Hospital, Antalya, Turkey (Türkiye)